CLINICAL TRIAL: NCT03260387
Title: Advancing Treatment for Pancreatitis: A Prospective Observational Study of TPIAT (POST)
Brief Title: A Prospective Observational Study of TPIAT
Acronym: POST
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Baylor Health Care System (Other); Medical University of South Carolina (Other); University of Chicago (Other); University of Pittsburgh Medical Center (Other); Dartmouth-Hitchcock Medical Center (Other); Johns Hopkins University (Other); Children's Hospital Medical Center, Cincinnati (Other); Ohio State University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: PEDS-2019-26517; R01DK109124 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pancreatitis, Chronic; Pancreatectomy; Hyperglycemia; Pancreatitis
Keywords: pediatric; total pancreatectomy; acute pancreatitis; chronic pancreatitis; islet transplant; islet autotransplant
MeSH Terms: conditions — Pancreatitis, Chronic; Hyperglycemia; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional (opt in) biorepository samples:
  1. Blood (plasma, serum, buffy coat)
  2. Urine
  3. Saliva
  4. Pancreas biopsy at time of surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TPIAT: patients undergoing total pancreatectomy with islet autotransplant.
  Interventions: Procedure: TPIAT

INTERVENTIONS:
Procedure: TPIAT — The entire pancreas is removed to treat the pain of chronic pancreatitis, and the islets are infused back into the patient to reduce diabetes risk after surgery.

SUMMARY:
Multi-center, prospective, observational cohort study of patients undergoing total pancreatectomy with islet autotransplantation (TPIAT)

DETAILED DESCRIPTION:
Patients who are undergoing TPIAT at one of the participating center are invited to participate in this observational study, with 450 participants anticipated. The aims of the study are:

Aim 1: To determine (1a) whether patient and disease characteristics are associated with favorable pain and health-related quality-of-life outcomes (HRQOL) after TPIAT; (1b) the optimal timing of the TPIAT intervention to resolve pain and improve HRQOL; and (1c) in a subset of patients, the impact of central sensitization on pain resolution.

Aim 2: To determine (2a) whether patient and disease characteristics are associated with favorable glycemic outcomes from the IAT procedure; and (2b) the optimal timing of TPIAT to obtain post-surgical insulin independence.

Aim 3: To determine the cost-effectiveness of TPIAT.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with chronic or recurrent acute pancreatitis undergoing total or completion pancreatectomy with islet autotransplantation at a participating center.

Exclusion Criteria:

1. Partial pancreatectomy
2. TPIAT performed for a diagnosis other than chronic or recurrent acute pancreatitis (for example benign or malignant pancreatic tumor)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and Adults undergoing TPIAT for severe pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Reduction | Mos 6, Years 1, 2, 3, 4 after surgery
  Visual Analog Pain Scale
Quality of Life | Mos 6, Years 1, 2, 3, 4 after surgery
  Physical Component Summary Score from SF-12
Quality of Life | Mos 6, Years 1, 2, 3, 4 after surgery
  Mental Component Summary Score from SF-12
Diabetes | Mos 6, Years 1, 2, 3, 4 after surgery
  Proportion of patients insulin independent

SECONDARY OUTCOMES:
Opioid Use | Mos 6, Years 1, 2, 3, 4 after surgery
  proportion off opioid analgesics
Opioid Use | Mos 6, Years 1, 2, 3, 4 after surgery
  Morphine Equivalents (avg daily ME)
Glycemic Control | Mos 6, Years 1, 2, 3, 4 after surgery
  HbA1c level
Insulin Dose | Mos 6, Years 1, 2, 3, 4 after surgery
  Insulin Dose (U/day)
Islet Graft Function | Mos 6, Years 1, 2, 3, 4 after surgery
  Proportion with Islet Graft Function (C-peptide + or Off Insulin)
Severe Hypoglycemia Episodes | Mos 6, Years 1, 2, 3, 4 after surgery
  Proportion of patients with Severe Hypoglycemia
Pain Interference | Mos 6, Years 1, 2, 3, 4 after surgery
  Pain interference Score (PROMIS scale)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of California, San Francisco, San Francisco, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Thomas E. Starzl Transplantation Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No